CLINICAL TRIAL: NCT01225458
Title: Behaviour and Cognitive Evaluation for Dialysis Elderly Patients (BCDE)
Acronym: BCDE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BCDE
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Renal Insufficiency; Chronic Kidney Failure; Aged
Keywords: Elderly patients; renal insufficiency; systematized gerontologic evaluation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- exclusive nephrology follow-up (Placebo Comparator): 250 patients will be included and randomized in the "exclusive nephrology follow-up" arm will continue their usual nephrology follow-up with consultations every 6 months during 3 years for dialysis patients or with consultations every 6 months before dialysis, 3 months after starting dialysis and every 6 months for a total duration of 3 years for non-dialysis patients. In addition to their nephrology consultations, patients will benefit from a geriatric evaluation with MMS, GDS and ADL scoring.
  Interventions: Other: shorter tests; Other: initial complete geriatric tests
- geriatric follow-up (Experimental): 250 patients will be included and randomized in the "geriatric follow-up" arm. They will continue their usual nephrology follow-up with consultations every 6 months during 3 years for dialysis patients or with consultations every 6 months before dialysis, 3 months after starting dialysis and every 6 months for a total duration of 3 years for non-dialysis patients.
  About geriatric evaluation Patients randomized in this arm will also have more complete tests to evaluate cognitive functions (memory, language and movements), psychological functions (depression and anxiety) and dependency in activities of daily living. Other tests will allow evaluate vision, audition, mobility and nutritional status.
  Interventions: Other: shorter tests; Other: initial complete geriatric tests; Other: follow-up complete geriatric tests

INTERVENTIONS:
Other: shorter tests — Geriatric evaluation with MMS, GDS and ADL scoring
Other: initial complete geriatric tests — evaluation of cognitive functions, psychological functions, dependency in activities, vision, audition, mobility and nutritional status : only at the first visit
Other: follow-up complete geriatric tests — evaluation of cognitive functions, psychological functions, dependency in activities, vision, audition, mobility and nutritional status : every 6 month for 3 years
  Arms: geriatric follow-up

SUMMARY:
The trial is a multicenter, prospective, randomized, open study. A total of 500 elderly patients aged over 75 years with renal insufficiency stage 5 will be included in the study after signed informed consent. Patients will be randomized 1/1 in two arms : 250 patients in the "exclusive nephrology follow-up" arm will continue their usual follow-up; 250 patients in the "geriatric follow-up" arm will have both their usual nephrology follow-up and a geriatric follow-up.

The aim of the study is to determine if a systematized gerontologist evaluation delay the occurrence of a composite primary endpoint : death, dementia, depression and severe dependency. The hypothesis is that the functional and vital prognosis of a patient with renal insufficiency depends not only on common and classical factors but also on cognitive and psychological functions and dependence, particularly in elderly patients.

ELIGIBILITY:
Inclusion criteria :

* Patients aged of 75 years old or more,
* Chronic kidney disease stage 5 defined by :
* either an estimated GFR (MDRD) ≤ 15ml/mn/1,73 m² in a non-dialysis patient with a nephrology follow-up > 3 months ("Pre-dialysis cohort"),
* or a dialysis treatment started for more than 3 months and less than one year, after a pre-dialysis follow-up > 3 months ("post-dialysis cohort"),
* Signed and dated informed consent.

Exclusion criteria :

* Moderately severe to severe dementia (MMS ≤ 15),
* Major depression and/or GDS-15 > 10/15,
* Severe dependency (ADL < 3/6).,
* Psychosis, mutism or aphasia,
* Malignancy or any pathology with life expectancy < one year.
* Ongoing specialized geriatric care

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
death | every 6 month for 3 years since inclusion
occurrence of a severe dementia (MMS < 10) | every 6 month for 3 years since inclusion
major depression detected by GDS-15 > 10/15 and confirmed by DSM-IV criteria | every 6 month for 3 years since inclusion
severe dependency (ADL < 3/6) | every 6 month for 3 years since inclusion

SECONDARY OUTCOMES:
cognitive, psychic and autonomy scores | every 6 month for 3 years since inclusion
cardiovascular morbidity and mortality | every 6 month for 3 years since inclusion
bone fracture | every 6 month for 3 years since inclusion
nutritional parameters | every 6 month for 3 years since inclusion
dialysis parameters | every 6 month for 3 years since inclusion
biological follow-up of chronic kidney disease including haemoglobin level | every 6 month for 3 years since inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France